CLINICAL TRIAL: NCT04518618
Title: The Effect of Adding Ultra-low Dose of Naloxone to Fentanyl on the Incidence of Pruritis After Spinal Anesthesia for Cesarean Section: Prospective Randomized Double-blind Study ÏÑÇÓÉ
Brief Title: Effect of Intrathecal Naloxone in the Incidence of Pruritis After C.S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Clinical Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 33954/7/20
Record Dates: First submitted 2020-08-11; First posted 2020-08-19 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Pruritis
Keywords: Pruritis; Naloxone; Spinal anesthesia; Fentanyl; Cesarean section
MeSH Terms: conditions — Pruritus | interventions — Fentanyl; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * The patients will be blinded to their groups.
  * An anesthesia resident who will not participate in the study and have no subsequent rule in it will help in the preparation of local anesthetic mixtures under strict aseptic precautions.
  * The anesthetist who will perform the spinal anesthesia will be blinded to the local anesthetic mixtures he will inject intrathecally.
  * An assistant nurse who will be blinded to the study groups and will have no subsequent rule in it will help in collection of the data of measurments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group F (Experimental): Patients in this group will receive spinal anesthesia with 10 mg hyperbaric bupivacaine (2 ml) plus 25 ugs of fentanyl (0.5 ml).
  Interventions: Drug: Fentanyl
- Group FN (Experimental): Patients in this group will receive spinal anesthesia with 10 mg hyperbaric bupivacaine (2 ml) plus 25 ugs of fentanyl (0.5 ml) plus 20 ugs naloxone.
  Interventions: Drug: Fentanyl; Drug: Naloxone

INTERVENTIONS:
Drug: Fentanyl — Spinal anesthesia will be performed with injection of 2.5 ml which will be composed of 10 mg hyperbaric bupivacaine (2 ml) and 25 ugs fentanyl (0.5 ml)
  Other Names: Intrathecal Fentanyl alone
Drug: Naloxone — Spinal anesthesia will be performed with injection of 2.5 ml which will be composed of 10 mg hyperbaric bupivacaine (2 ml) and fentanyl 25 ug combined with 20 ugs naloxone in 0.5 ml
  Other Names: Intrathecal fentanyl and naloxone
  Arms: Group FN

SUMMARY:
This randomized prospective double-blind trial will be conducted on 80 Full-term pregnant females aged 21- 30 years presented for elective cesarean section under spinal anesthesia where they will be randomly allocated into two equal groups:-

* Group F (40 Patients): Patients in this group will receive spinal anesthesia with 10 mg hyperbaric bupivacaine (2 ml) plus 25 ug of fentanyl (0.5 ml).
* Group FN (40 patients): Patients in this group will receive spinal anesthesia with 10 mg hyperbaric bupivacaine (2 ml) plus 25 ug of fentanyl (0.5 ml) plus 20 ug naloxone.

The study aim is to evaluate the effect of adding an ultra-low dose of naloxone (20 ug) to hyperbaric bupivacaine (10 mg0 and fentanyl (25 ug) in spinal anesthesia for C.S.

Primary outcome: The incidence of pruritis Secondary outcome: The onset, the duration, the site, and the severity of pruritis.

DETAILED DESCRIPTION:
This prospective randomized double-blind study will be carried out on 80 female patients who will be presented for elective C.S in the Obstetric department in Tanta university hospitals.

Full-term pregnant female aged 21- 30 years presented for elective cesarean section under spinal anesthesia will be included in the study.

The patients will be randomly allocated into two groups by the aid of computer-generated software of randomization. All the local anesthetic mixtures will be prepared under complete aseptic precautions by an anesthesia resident who will not participate in the study and will be blinded to its groups in to: - Group F (40 Patients): Patients in this group will receive spinal anesthesia with 10 mg hyperbaric bupivacaine (2 ml) plus 25 ug of fentanyl (0.5 ml).

Group FN (40 patients): Patients in this group will receive spinal anesthesia with 10 mg hyperbaric bupivacaine (2 ml) plus 25 ug of fentanyl (0.5 ml) plus 20 ugs naloxone.

Once the patient will be admitted to the operating theatre, all monitors will be applied with introduction of 18-gauge peripheral venous cannula and starting fluid preload in the form of lactated ringer solution 7 ml/kg over 30 minutes. While the patient in a sitting position and under complete aseptic precautions, patients will receive spinal block at lumbar 3-4 or 4-5 intervertebral space with an injection of the pre-prepared local anesthetic mixture according to the group of patient. After giving anesthesia and positioning for surgery with a left lateral tilt of 15 degrees, supplemental oxygen at a rate of 4 liters/minute will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Full-term pregnant female aged 21- 30 years presented for elective cesarean section under spinal anesthesia.

Exclusion Criteria:

* Patients with pregnancy less than 36 weeks or more than 40 weeks
* Patients with hypertension, pre-eclampsia, or eclampsia.
* Patients with diabetes
* Patients with cardiovascular disease and /or arrhythmia.
* Patients with placenta previa, accreta, percreta.
* Obese patients with BMI >36 Kg/m2
* Patients with height less than 160 Cm
* Multigravida
* Polyhydramnious patients

Ages: 21 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Full-term pregnant females undergoing elective C.S
Enrollment: 96 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
The incidence of pruritis | The first 24 hours postoperatively
  The percent of patients who will complain from pruritis in the first 24 hours after surgery

SECONDARY OUTCOMES:
The onset of pruritis | through study completion, average 4 months
  The time interval in minutes from the intrathecal injection to the first incidence of pruritis
The duration of pruritis | through study completion, average 4 months
  the time interval from the first incidence to the last incidence of pruritis
The Severity of pruritis | through study completion, average 4 months
  pruritis VAS score (PVAS is a 10cm long line and a single question, it is most commonly used in clinical trials for measuring itch intensity and features high reliability and concurrent validity. The left end point represents gno itch h and the right end point the gworst imaginable itch). It can be interpreted as follows: VAS 0= No pruritus, VAS < 3 = Mild pruritus, VAS 3-6 = Moderate pruritus, VAS 7-8 = Severe pruritus, VAS . 9=Very severe pruritus.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelkhalik, M.D, Principal Investigator — Tanta University
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Tanta, Algharbia
  - Tanta University hospitals, Tanta

IPD SHARING:
Plan to Share IPD: Yes
The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Supporting Information: SAP, ICF
Time Frame: 6 months after approval of the publication of the trial.
Access Criteria: Contact the principle investigator